CLINICAL TRIAL: NCT03010566
Title: Studying the Microbiome of the Lung in Patients Treated With Endobronchial Lung Volume Reduction Coils for Emphysema
Brief Title: Lung Volume Reduction Coil Microbiome Study
Acronym: LVRC-Micro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 215696
Record Dates: First submitted 2016-12-20; First posted 2017-01-05 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
Keywords: Lung volume reduction coil; Lung Microbiome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oropharyngeal swab, Broncho-alveolar lavage, Bronchial brushings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studying the microbiome of the lung in patients treated with endobronchial lung volume reduction coils for emphysema

DETAILED DESCRIPTION:
Patients with severe emphysema and hyperinflation can benefit from lung volume reduction techniques designed to reduce gas trapping, improve air flow, and restore more natural chest wall and lung mechanics. The best evidence exists for lung volume reduction surgery (LVRS), but more recently there has been increasing interest in, and use of, bronchoscopic lung volume reduction (BLVR) techniques. One of the more intriguing methods has been the use of endobronchial lung volume reduction coils (LVRCs), nitinol wires which when deployed in the lung take up their preformed shape similar to that of a tennis ball seam, and seem to work both by mechanical compression of lung tissue and by replacing some of the elastic recoil forces that are lost when there is emphysematous destruction of lung tissue. Treatment aims to place 10 coils in each upper lobe in 2 procedures separated by 1-3 months.

A number of studies on the use of LVRCs have now been published, but most of these provide only relatively short term follow-up and safety data. Fairly widespread clinical use of the LVRC is now occurring in Germany, however. It is now being increasingly recognised that a minority of patients treated with LVRCs (approximately 5-10%) develop dense consolidation around one or more of their devices, with the development of significant cavitation in some of these patients. At least 1 death has been attributed to decline associated with the development of such changes, and a number of other patients have now developed infection with persistent and resistant organisms. Unlike endobronchial valves (currently the most widely used of the BLVR devices), patients are told that LVRC treatment is permanent and that the devices cannot be removed after implantation, something which obviously has implications if devices become infected or colonised with micro-organisms.

The lung microbiome is the complete collection of microorganisms that inhabit the lung, including bacteria, viruses, and fungi. Studies have demonstrated the importance of microorganisms in the pathogenesis of chronic obstructive pulmonary disease (COPD), and in driving exacerbations and loss of lung function, and the lungs of patients with severe COPD (those potentially suitable for LVRC treatment) contain a different community of bacteria to those of healthy people. Culture-independent molecular techniques are now available for precise cataloguing of the lung microbiome, with results that are far more detailed and informative than standard culture techniques. By DNA sequencing the 16S rRNA gene and using it as a barcode to identify all bacterial organisms in any given sample and also their relative proportions, a much broader, less selective group of bacteria can be assayed.

The bilateral sequential nature of LVRC treatment provides a unique opportunity for the collection of multiple samples from each patient at different time points in their treatment, and thus to track changes in the lung microbiome that may be caused by LVRC implantation. It is now our practice to perform a bronchoscopy 6 months after initial treatment in all patients who have undergone BLVR (LVRCs, endobronchial valves, thermal vapour ablation) in order to monitor for device migration, granulation tissue formation, and to obtain specimens for bacterial culture. This therefore means that LVRC patients undergo bronchoscopy on 3 occasions, spaced approximately 3 months apart.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for lung volume reduction coil treatment for the management of severe emphysema

Exclusion Criteria:

* Unwilling or unable to sign the informed consent form
* Patients with known Category 3 Organisms as per the Advisory Committee on Dangerous Pathogens (ACDP) for example, Tuberculosis or Human Immunodeficiency Virus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe emphysema who are scheduled to undergo endobronchial lung volume reduction coils insertion
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in the microbiome of the lungs in patients treated with lung volume reduction coils (LVRCs). | 6 months

SECONDARY OUTCOMES:
Correlation between signals from 16S rRNA gene-sequencing analysis at baseline and infective complications following LVRC treatment. | 6 months
Genome sequencing of dominant pathogens to determine virulence factors. | 6 months
Genome sequencing of dominant pathogens to determine antibiotic resistance. | 6 months
Genome sequencing of dominant pathogens for strain-level identification. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel V Kemp, MBBS MD, Principal Investigator — Royal Brompton & Harefields Hospital
Locations (2):
- United Kingdom (2):
  - Chelsea & Westminster Hospital, London, Chelsea
  - Royal Brompton & Harefields Hospital, London, Fulham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kozich JJ, Westcott SL, Baxter NT, Highlander SK, Schloss PD. Development of a dual-index sequencing strategy and curation pipeline for analyzing amplicon sequence data on the MiSeq Illumina sequencing platform. Appl Environ Microbiol. 2013 Sep;79(17):5112-20. doi: 10.1128/AEM.01043-13. Epub 2013 Jun 21. PMID 23793624